CLINICAL TRIAL: NCT06951919
Title: HOme-Based Self-management and COgnitive Training CHanges Lives (HOBSCOTCH) - Multiple Sclerosis (MS) - Efficacy Trial
Brief Title: HOBSCOTCH-MS-Efficacy Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Elaine T. Kiriakopoulos, MD, MPH, MSc Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02002897
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Cognitive Dysfunction; Memory Disorders; Memory Impairment; Memory Dysfunction
Keywords: Cognition; Self-Management; Cognitive Remediation; Cognitive Training; Memory Disorders; Caregivers; Caregiver Burden; Mindfulness
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Memory Disorders; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MS Participant Group 1 (Experimental): MS Participant Group 1 will receive the HOBSCOTCH-MS intervention consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH
  * Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: Home Based Self- management and Cognitive Training Changes lives in Multiple Sclerosis (HOBSCOTCH-MS)
- MS Participant Group 2 (Active Comparator): MS Participant Group 2 will be on a 3-month wait list after which they will receive HOBSCOTCH-MS consisting of 1:1 sessions delivered once per week including:
  * 1 pre-HOBSCOTCH
  * Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions
  * 1 wrap-up session (webcam or telephone)
  Interventions: Behavioral: Home Based Self- management and Cognitive Training Changes lives in Multiple Sclerosis (HOBSCOTCH-MS)
- MS Caregiver Group 1 (Experimental): Caregiver Group 1 will receive an adapted version of HOBSCOTCH-MS by attending the introductory session and session 1 of the HOBSCOTCH-MS (virtual) program with their MS participant as well as guidance and instructions on utilizing quick relaxation. Caregiver Group 1 will also attend session 8 of the program with the MS patient to focus on program wrap-up and maintenance planning.
  Interventions: Behavioral: Home Based Self- management and Cognitive Training Changes lives in Multiple Sclerosis (HOBSCOTCH-MS)
- MS Caregiver Group 2 (Active Comparator): Caregiver Group 2 will be on a 3 month wait list with their MS participant after which time they will receive an adapted version of HOBSCOTCH-MS by attending the introductory session and session 1 of the HOBSCOTCH-MS (virtual) program with their MS patient as well as guidance and instructions on utilizing quick relaxation. Caregiver Group 1 will also attend session 8 of the program with the MS patient to focus on program wrap-up and maintenance planning.
  Interventions: Behavioral: Home Based Self- management and Cognitive Training Changes lives in Multiple Sclerosis (HOBSCOTCH-MS)

INTERVENTIONS:
Behavioral: Home Based Self- management and Cognitive Training Changes lives in Multiple Sclerosis (HOBSCOTCH-MS) — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-MS is an adaptation of the HOBSCOTCH program specifically for people who have multiple sclerosis. It incorporates education about these conditions and cognition into the education module.
  Other Names: HOBSCOTCH-MS

SUMMARY:
The purpose of this study is to assess the ability of the home-based intervention, HOBSCOTCH-MS to improve the quality of life and cognitive function in Service Members, Veterans and civilians who have multiple sclerosis with cognitive and memory problems (MS participants). This study will also assess the ability of the HOBSCOTCH-MS program to improve quality of life in caregivers of patients with multiple sclerosis and to reduce caregiver burden. Enrolling with a Caregiver is optional for MS participants.

Investigators will compare two groups of MS participants and their Caregiver (enrolling with a Caregiver is optional): one who receives HOBSCOTCH-MS immediately (Group 1) and another group that will receive HOBSCOTCH-MS (Group 2) after a 3-month waiting period. Participants will be in the study for about 6 months total.

HOBSCOTCH-MS involves 45 to 60 minute one on one virtual sessions with a certified Cognitive Coach including a "pre" program session and 8 weekly sessions thereafter. Participants will learn about problem solving therapy and mindfulness or relaxation training. MS participants are asked to do short homework assignments and both MS and Caregiver participants are asked to keep a brief daily diary on a smart phone app. All participants complete study questionnaires or surveys at enrollment, 3 months later and at 6 months (at the end of the study).

After completing the intervention, MS Participants and their Caregivers may also participate in an optional one-time Key Informant Interview for qualitative analysis in an effort to further adapt and improve the HOBSCOTCH-MS in the future.

DETAILED DESCRIPTION:
The investigators' hypothesis is that the telehealth delivered evidence-based intervention HOBSCOTCH-MS can be delivered by telehealth to improve QOL and neurocognitive function in PwMS. The innovative integration of care partner participation in the proposed coproduced adapted intervention, HOBSCOTCH-MS, will reduce care partner burden and increase care partner knowledge of their loved one's disease and the cognitive challenges they face, leading to an improvement in care partner QOL.

SPECIFIC AIMS: The investigators will test their hypothesis by pursuing the following specific aims:

Aim 1. Evaluate the efficacy of HOBSCOTCH-MS in persons with MS. The investigators' working hypothesis is that treatment will be associated with gains in QOL and subjective cognition in people with multiple sclerosis. The investigators also expect to see improvements in problem-solving ability, objective cognition, knowledge, self-efficacy, and mood. We will examine predictors of response to treatment, including baseline cognition, mood, fatigue, and demographic and disease variables, and mediators including problem-solving abilities and self-efficacy.

Aim 2. Evaluate the efficacy of HOBSCOTCH-MS in care partners (caregivers). The investigators' working hypothesis is that care partners (caregivers) will have improvement in health-related QOL, care partner burden, knowledge, self-efficacy, and mood as a result of their family member with MS participating in the intervention, and by their own participation in education and mindfulness exercises.

Aim 3: Collect and synthesize key informant interview data from a subset of participating people with multiple sclerosis (MS participants) and their Care Partners (Caregiver participants) to inform a future larger scale trial. The investigators' working hypothesis is this qualitative data will assist with refinements to materials and/or program delivery that would recognize and validate key input from people with multiple sclerosis and their care partners (caregivers), allowing the investigators to plan for future large scale research trials and program dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - MS Participant

  * Age 20 - 75 years
  * Diagnosis of relapsing or progressive MS
  * Education of at least Grade 12 or GED
  * Fluent in English
  * Subjective cognitive and memory challenges
  * Internet access
  * Telephone access

Inclusion Criteria - Caregiver Participant

* 20 years +
* Fluent in English
* Caregiver to a MS Participant
* Participant MS has given permission to Caregiver to enroll with them
* Internet access
* Telephone access

Exclusion Criteria:

* Exclusion Criteria MS Participant

  * Current diagnosed psychiatric disorders (e.g., schizophrenia, bipolar disorder or substance use disorder).
  * Other neurological disorder such as epilepsy, brain tumor, severe brain injury or mild to moderate brain injury with a history of 30 or more minutes' loss of consciousness, or other disorder that would confound the focus on MS
  * Diagnosed developmental attention, learning, or intellectual disorder; sensory, motor, or physical disability that would prevent engagement with the intervention or render the person unable complete study outcome measures
  * Exacerbation of MS symptoms (relapse) or ongoing steroid treatment within three months of study enrollment
  * Significant visual impairment precluding reading or writing
  * Lack of access to the technical resources (e.g., internet access, telephone) required for participation

Exclusion Criteria - Caregiver Participant

* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life in MS participants as measured by comparing PROMIS-10 Global Health scores at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention
  PROMIS Global-10 Global Health is a validated 10-question survey and part of the Patient-Reported Outcomes Measurement Information System (PROMIS) used to assess health care-related quality of life. Measures include overall health, pain, fatigue, social health, mental health, and physical health. 9 of the items are scored on a Likert Scale of 1 - 5 with 5 representing the best health care-related quality of life; higher scores are associated with better quality of life. One item related to pain is measured on a scale of 1 - 10 with 10 being the worst possible pain.
Change in subjective cognitive function in MS participants as measured by comparing scores on the Cognitive Function Sub-Scale (Item Bank 2.0) of the Neuro-QOL at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Change in Caregiver participants caregiver burden as measured by comparing Zarit Burden Interview scores at baseline and at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5 point Likert scale is used with a higher score indicating a greater level of perceived burden.

SECONDARY OUTCOMES:
Changes in MS and Caregiver participants' knowledge of relationship between the condition of MS and cognition and memory as measured by comparing scores on the HOBSCOTCH-MS Knowledge Questionnaire at baseline and at 6 months (end of study). | Baseline and at 6 months (end of study)
  The MS Knowledge Questionnaire is a 12-item Yes/No (true/false) questionnaire that was developed by the study team at the HOBSCOTCH Institute. It is scored based on number of correct responses.
Change in MS participants quality of life as measured by comparing FAMS-Functional Assessment of Multiple Sclerosis v4.0 scores at base line and at 3 months post-HOBSCOTCH-MS intervention. | Baseline and 3 months post-intervention
  The Functional Assessment of Multiple Sclerosis (FAMS) is a validated self-report health-related quality-of-life instrument for people with multiple sclerosis. The FAMS consists of 44 scored (5-point Likert scale) items in six quality-of-life domains: Mobility (seven items), Symptoms (seven items), Emotional wellbeing (seven items), General contentment (seven items), Thinking/fatigue (nine items), and Family/social wellbeing (seven items). An Additional concerns subscale consists of 15 other items that fall outside of the six domains but may provide valuable information to the clinician. The FAMS includes items across the International Classification of Functioning components of body functions, activities and participation, and environmental factors. Higher scores indicate better quality of life.
Change in MS participants objective cognitive processing speed as measured by comparing Symbol-Digit Modalities Test scores (orally) at base line and at 3 months post-HOBSCOTCH-MS intervention. | Baseline and 3 months post-intervention
  The Symbol Digit Modalities Test (SDMT) is a validated tool that objectively measures cognitive processing speed. It requires a person to substitute a number (1 - 9), either orally or written, for randomized presentations of geometric figures over 90 seconds. Scores range between 0 and 100 with a lower score representing poorer performance.
Change in MS participants verbal learning and memory as measured by comparing California Verbal Learning Test-III scores at baseline and 3 months post-HOBSCOTCH-MS intervention | Baseline and 3 months post-intervention
  The California Verbal Learning Test-III is an objective, validated verbal learning and memory assessment. It consists of a 16-word, list-recall task with up to five learning/recall trials. Higher scores of recall over time are associated with better performance.
Change in MS participants visuospatial learning and memory as measured by comparting Brief Visuospatial Memory Test-Revised (BVMT-R) scores at baseline and 3 months post-HOBSCOTCH-MS intervention | Baseline and 3 months post-intervention
  The Brief Visuospatial Memory Test - Revised (BVMT-R) is an objective, standardized assessment to measure visuospatial learning and memory abilities. It consists of six equivalent, alternate BVMT-R stimulus forms of six geometric figures printed in a 2 x 3 array on a separate page of the Recall Stimulus Booklet. In the three Learning Trials, the respondent views the Recall Stimulus page for ten seconds and then is asked to draw as many of the figures as possible in their correct location on a page in the Response Booklet. After a 25-minute delay which includes primarily verbal activities, the task is repeated. Then, the respondent is asked to identify which of the 12 figures in the Recognition Stimulus Booklet were included in the six geometric figures on the original Recall Stimulus page. Higher scores on each of the three trials represent better visuospatial learning and memory.
Changes in MS participants executive function as measured by comparing scores on the self-reported Behavior Inventory of Executive Function-Adult Version (BRIEF-A) at baseline and 3-months post intervention. | Baseline and 3 months post-intervention
  The BRIEF-A is a standardized measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment that includes 75 items within nine scales of executive function. All 75 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). Raw scores for each scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores indicate greater impairment in executive functioning.
Changes in MS participants self-efficacy as measured by comparing scores on the PROMIS (Patient-Reported Outcomes Measurement Information System) Item Bank v1.0 General Self-Efficacy assessment at baseline and 3-months post-intervention. | Baseline and 3 months post-intervention
  The PROMIS self-efficacy scales is a validated measure designed to assess an individual's confidence in managing various situations, problems and events. 10 items are self-reported on a scale of 1 (I am not at all confident) to 5 (I am very confident). Lower scores indicate poorer perception of self-efficacy.
Changes in MS participants and Caregiver participants mood as measured by comparing scores on the Patient Health Questionnaire (PHQ-9) at baseline and at 3 months post- intervention. | Baseline and 3 months post-intervention
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria on a 4-point Likert scale as "0" (not at all) to "3" (nearly every day). Higher scores are consistent with greater symptoms of poor mood or depression.
Changes in MS participants and Caregiver participants anxiety as measured by comparing score on the Generalized Anxiety Disorder-7 (GAD-7) at baseline and at 3-months post-intervention. | Baseline and 3 months post-intervention
  The Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring symptoms of generalized anxiety disorder (GAD). The seven items are scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Higher scores suggest greater symptoms of anxiety.
Changes in MS participants' symptom frequency as measured by a daily self-reported diary compared at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention
  MS participants will self-report by checking off any of 10 common MS symptoms using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in MS participants' medication adherence as measured by a daily self-reported diary of compared at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention
  MS participants will self-report their medication adherence activity using a smartphone app or paper log checking yes/no to taking medications that day. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in MS participants' use of memory strategies as measured by a daily self-reported diary compared at baseline and 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention
  MS participants will self-report their use of the memory strategies they learn in the HOBSCOTCH-MS program by checking yes/no using a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in a paper log.
Changes in Caregiver participants use of quick relaxation strategies as measured by a daily self-reported diary compared at baseline and 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention
  Caregiver participants will self-report their use of the quick relaxation strategies they learn in the HOBSCOTCH-MS program by checking yes/no using a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in a paper log.
Changes in MS participants and MS Caregiver participants self-reports of wellbeing as measured by comparing daily reports of well-being in a diary at baseline and at 3 months post-intervention. | Recorded daily and compared between baseline and 3 months post-intervention
  MS participants and Caregiver participants will self-report daily well-being information throughout the entire study by use of a smartphone app or paper log and a basic 5-item item Likert-scale of well-being ranging from Very Poor to Great.
Engagement and Satisfaction for MS participants as measured by analyzing study attrition and a Participant Satisfaction Survey at the end of the study. | At 6 months (end of study participation)
  The Participant Satisfaction Survey has been developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It contains 10 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program.
Engagement and Satisfaction for MS Participants as measured by CollaboRATE post-study completion. | At 6 months (end of study participation).
  CollaboRATE is a brief, 3 item patient-reported measure of shared decision making, namely the perception of being informed and then involved in decision-making steps. A 10-point anchor scale from 0 (no effort was made) to 9 (every effort was made) with higher scores representing a greater perception of a shared decision-making effort.
HOBSCOTCH-MS fidelity as measured by MS participant's compliance with weekly homework assignments. | Week 1 through Week 8 of HOBSCOTCH-MS intervention.
  Homework assignments are given each week in which participants are asked to think about solutions using the Problem Solving Therapy taught in the program. Compliance is measured by Yes (completed homework assignment) or No (did not complete homework assignment).
Changes in MS Caregiver participants self-reported health status as measured by comparing scores on the Short-Form Health Survey 36 (SF-36) at baseline and 3 months-post HOBSCOTCH MS intervention. | Baseline and 3 months post-intervention
  The Short Form Health Survey (SF-36) is a validated 36-item, patient- reported survey of patient health. It consists of 8 sub-scales, which are scored on a 3-point, 5-point or dichotomous (yes/no or true/false) scale. The scores are converted to a 1 - 100-point scale with a lower score indicating more disability, i.e. 0 = maximum disability and 100 = no disability.
Feasibility of HOBSCOTCH-MS program for Caregivers as measured by study attrition and a Participant Satisfaction Survey. | At 6 months (end of study participation)
  The Participant Satisfaction Survey was developed through the original HOBSCOTH program and is used in clinical practice for quality improvement. It has been modified to address Caregiver's satisfaction as a result or participating in this study and contains 9 items scored on a 5- point Likert scale with a higher score indicating greater satisfaction with the program.
Sustainability of improvement on primary outcome measure of quality of life for Group 1 MS Participants by comparing scores on the PROMIS 10-Global Health at 3 months and 6 months post-intervention. | 3 months and 6 months post intervention
  PROMIS Global-10 Global Health is a validated 10-question survey and part of the Patient-Reported Outcomes Measurement Information System (PROMIS) used to assess health care-related quality of life. Measures include overall health, pain, fatigue, social health, mental health, and physical health. 9 of the items are scored on a Likert Scale of 1 - 5 with 5 representing the best health care-related quality of life; higher scores are associated with better quality of life. One item related to pain is measured on a scale of 1 - 10 with 10 being the worst possible pain.
Sustainability of improvement on primary outcome measure of quality of life for Group 1 MS Participants by comparing scores on the Neuro-QOL at 3 months and 6 months post-intervention. | 3 months and 6 months post intervention
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.
Sustainability of improvement on primary outcome measures for Group 1 Caregiver Participants by comparing scores on the Zarit Caregiver Burden at 3 months and 6 months post-intervention. | 3 months and 6 months post intervention
  The Zarit Burden Interview is a 22-item questionnaire designed to measure the extent to which a caregiver perceives his or her level of burden as a result of caring for a person with a particular diagnosis. A 5-point Likert scale is used with a higher score indicating a greater level of perceived burden.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, Principal Investigator — Dartmouth-Health/Dartmouth-Hitchcock, Dartmouth College
Locations (1):
- Dartmouth-Health Lebanon, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No